CLINICAL TRIAL: NCT07065669
Title: Treating Adolescent Obsessive Compulsive Disorder With Transcranial Magnetic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Hearst Foundations (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-41216
Record Dates: First submitted 2025-06-23; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Adolescent; transcranial magnetic stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Two arm, randomized assignment to two types of transcranial magnetic stimulation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Right Orbitofrontal TBS (Experimental): continuous theta burst stimulation
  Interventions: Device: cTBS to ROFC
- TBS of dorsal, medial prefrontal cortex (Active Comparator): intermittent theta burst stimulation (iTBS) will be delivered to the dmPFC
  Interventions: Device: Dorsal medial Prefrontal Cortex intermittent theta burst stimulation

INTERVENTIONS:
Device: Dorsal medial Prefrontal Cortex intermittent theta burst stimulation — iTBS stimulation of the dmPFC is a FDA-approved treatment for adults with OCD
  Arms: TBS of dorsal, medial prefrontal cortex
Device: cTBS to ROFC — continuous theta burst stimulation (cTBS) 1,800 pulses per session
  Arms: Right Orbitofrontal TBS

SUMMARY:
This is a pilot study to examine the tolerability, safety and early efficacy of two forms of transcranial magnetic stimulation (TMS) for treating adolescents with Obsessive Compulsive Disorder (OCD) who have experienced limited improvements with usual treatments for OCD in adolescents.

The project's primary goal is to examine whether adolescents can complete 3 consecutive weeks of TMS administered 5 days per week, and to describe the type of and how common individual side effects with TMS occur in adolescents with OCD.

Participants will:

* visit the clinic every weekday for 3 weeks (15 days) to receive TMS treatments
* have a brain MRI scan before TMS treatments begins and after finishing all TMS
* complete questionnaires and report changes in behavior and physical symptoms

DETAILED DESCRIPTION:
This study's primary goal is to examine whether treatment with two forms of transcranial magnetic stimulation (TMS) called theta burst stimulation (TBS) show acceptable tolerability, safety, and preliminary signals of efficacy for adolescents with Obsessive Compulsive Disorder (OCD) that has not responded satisfactorily to 1st line treatments. While TMS is FDA-approved for OCD in adults, data on TMS in youth with OCD is limited. Results will inform on how suitable TMS treatment is for adolescents with OCD, and guide future, larger studies.

The study is considered a randomized, single blind, clinical trial.

The design of the study is a two-group parallel comparative study of two different TMS stimulation sites, the orbito-frontal cortex (OFC) and the dorsal medial prefrontal cortex (dmPFC).

Model description: both groups will receive active TMS treatment sessions in clinic every weekday for 3 consecutive weeks (15 days). During each TMS session, participants in both groups will receive 3 TMS stimulations separated by a rest period, for a total of 45 individual TMS treatments. Study participants will receive TMS to only their assigned stimulation site.

Number of arms: there are two treatment arms based on assigned treatment site, an OFC arm and a dmPFC arm.

Masking: an independent evaluator will be masked to treatment arm assignment and adverse events. All other study personnel will not be masked.

Allocation: participants will be randomly assigned to group according to a computer-generated assignment schedule.

Enrollment: total planned enrollment is 30 eligible participants who are randomized.

Arm Information:

Arm titles-- orbitofrontal cortex (OFC) and dorsal medial prefrontal cortex (dmPFC) Arm types: the dmPFC arm is considered the intervention arm; the OFC arm is considered the active comparator arm.

Interventions:

Intervention type: Device (both arms)

Intervention name(s):

OFC - continuous theta burst stimulation (cTBS) dmPFC - intermittent theta burst stimulation (iTBS)

Intervention description:

OFC - three stimulations per day of 1,800 pulses/stimulation cTBS for 15 days dmPFC - three stimulations per day of 1,800 pulses/session iTBS for 15 days

ELIGIBILITY:
Inclusion Criteria:

1. outpatients
2. ages 13 - 17 years
3. meets current DSM-5 criteria for Obsessive Compulsive Disorder with screening CY-BOCS II score > 16 (moderate to severe).
4. stable on chronic psychotropic medications and/or therapy for 8 weeks prior to the study and agreeable to continue throughout the study without changes.
5. participants may continue to take medications and record daily usage throughout the study.
6. capacity to provide informed assent and parent or legal guardian able to provide consent.
7. ability to tolerate clinical study procedures.
8. successfully complete the screening forms without any contraindications.

Exclusion Criteria:

1. Psychiatric: history of schizophrenia, bipolar disorder, substance/alcohol abuse disorder, current elevated suicide risk, prior psychosurgery, prior ECT.
2. Neurologic: severe neurocognitive disorder, seizure disorder, certain structural brain lesions (e.g., intracranial mass lesions, hydrocephalus, sequelae of meningitis, frank brain injury).
3. TMS contraindications: implanted device; presence of metal in the head, including eyes and ears (excluding dental implants); certain tics; medications or systemic illness that predispose seizure risk; family history of 1st degree relative with seizure disorder.
4. Subjects with an unstable physical, systemic, or metabolic disorder (e.g., unstable hypertension, malnutrition secondary to eating disorder).
5. Females who are pregnant or nursing (as determined by a questionnaire and pregnancy test).
6. Current and anticipated continued treatment with excluded medication (See prohibited list).
7. Inability to complete the research protocol as determined by the Principal Investigator.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Completion rate | Baseline to completion of all protocol visits, up to 8 weeks
  Proportion (percentage) of all participants who enter the study, undergo a minimum of one TMS treatment, and complete the protocol-specified 15 TMS visits
Adverse events | Baseline to completion of all protocol visits up to 8 weeks
  Frequency (percentage) of individual adverse events

SECONDARY OUTCOMES:
Combined efficacy | Baseline to completion of all protocol visits, up to 8 weeks
  Change in independent assessor-rated CY-BOCS II total score
Site efficacy | From screening to end of treatment (Week 4)
  Compare changes in blinded clinician CY-BOCS II total by TMS site (OFC vs dmPFC)

CONTACTS AND LOCATIONS:
Overall Officials: James T McCracken, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared will include both primary endpoint data and secondary endpoint data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning one year and ending 3 years after publication of results
Access Criteria: Qualified researchers who submit a brief description of planned analyses must be submitted to the PI to review and approve data sharing

REFERENCES:
- [Background] Vicheva P, Osborne C, Krieg SM, Ahmadi R, Shotbolt P. Transcranial magnetic stimulation for obsessive-compulsive disorder and post-traumatic stress disorder: A comprehensive systematic review and analysis of therapeutic benefits, cortical targets, and psychopathophysiological mechanisms. Prog Neuropsychopharmacol Biol Psychiatry. 2025 Jan 10;136:111147. doi: 10.1016/j.pnpbp.2024.111147. Epub 2024 Sep 16. PMID 39293504
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199